CLINICAL TRIAL: NCT05245851
Title: Clinical Deployment and Validation of Rho - An Opportunistic Osteoporosis Screening Software-as-a-Medical Device
Brief Title: Clinical Deployment and Validation of Rho
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 16 Bit Inc. (Industry)
Collaborators: Amgen (Industry); Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Rho_Pilot_PPV_341462
Record Dates: First submitted 2022-02-09; First posted 2022-02-18 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Low Bone Density
Keywords: osteoporosis; opportunistic; radiography; DXA
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis

STUDY DESIGN:
Intervention Model Description: 16 Bit intends to study the impact of RhoTM by performing a prospective trial to assess its impact. A selected pilot site must have both x-ray and dual energy x-ray absorptiometry (DXA) imaging services, with the anticipation that DXA referrals will be made to the same imaging center which performed the x-ray which underwent RhoTM screening. The study population to assess the impact of RhoTM will consist of patients aged 50 and above who are opportunistically screened by RhoTM while undergoing an x-ray of the lumbar spine, thoracic spine, hand, knee, pelvis or chest.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Opportunistic screening for low BMD (Experimental): Outpatients aged over 50 years undergoing x-ray of the thoracic spine, lumbar spine, chest, pelvis, hand or knee will have their x-rays screened for low BMD by the software-as-a-medical device. If low BMD is identified by the software, a radiologist reviewing the x-ray may choose to incorporate this as an incidental finding in their report to the referring physician.
  Interventions: Device: Opportunistic screening for low BMD

INTERVENTIONS:
Device: Opportunistic screening for low BMD — Software will analyze x-rays of the chest, thoracic spine, lumbar spine, pelvis, knee or hand/wrist acquired for any reason, and notify the radiologist at time of acquisition if low BMD is detected. The report to the radiologist includes the following statements:
  * This x-ray was opportunistically analyzed by RhoTM, an investigational device under ITA [investigational testing authorization] from Health Canada, to screen for low bone mineral density (low BMD).
  * This information should be used by a trained healthcare provider in conjunction with a patient's clinical fracture risk to determine if formal BMD screening with DXA is appropriate.
  The radiologist can choose to include this as an incidental finding in their report to the referring physician.

SUMMARY:
Osteoporosis is a widespread disease characterized by the loss of bone mineral density (BMD). 16 Bit has developed software, called RhoTM, that analyzes various x-rays, performed in patient age 50 and above for any clinical indication, to identify patients with low BMD. RhoTM is intended to function as a pre-screening device for low BMD. This study seeks to assess the clinical performance and impact of implementing RhoTM in real-world settings by analyzing its performance and impact on DXA referrals.

DETAILED DESCRIPTION:
Osteoporosis is a widespread disease characterized by the loss of bone mineral density (BMD). 16 Bit has developed an opportunistic screening tool for low BMD, called RhoTM, that analyzes lumbar spine, thoracic spine, chest, pelvis, knee, and hand radiographs, performed in patient age 50 and above for any clinical indication to estimate lumbar and femoral neck BMD. The estimated BMD T-score is used to classify patients as having normal or low BMD. A finding of low BMD can be included in a radiologist's report, and is intended to support a discussion between healthcare provider and patient regarding the need for osteoporosis diagnosis by dual-energy x-ray absorptiometry (DXA). In this way, RhoTM is intended to function as an opportunistic pre-screening device for low BMD. This study seeks to assess the clinical performance and impact of implementing RhoTM in real-world settings by analyzing the diagnostic performance and impact on DXA referrals.

ELIGIBILITY:
Inclusion Criteria:

* age 50+ years
* outpatient undergoing x-ray examinations of:
* chest
* thoracic spine
* lumbar spine
* pelvis
* knee
* hand/wrist

Exclusion Criteria:

* age < 50 years
* inpatient

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1146 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Positive predictive value | 9 months
  To measure the positive screening rate for all patients screened by RhoTM and the positive predictive value (PPV) in those patients who screen positive by RhoTM and undergo follow-up DXA. PPV will be assessed for identification of low BMD (T-score <-1) and for identification of moderate/high fracture risk.

SECONDARY OUTCOMES:
DXA conversion | 9 months
  To assess the DXA conversion rate defined as the proportion of patients who have a DXA within 6 months following a positively reported RhoTM screen. Scheduled DXA examinations may be used as a surrogate.

OTHER OUTCOMES:
Radiologist adoption | 2 months
  To assess radiologist adoption rate defined as the number of patients who are screened positive by RhoTM and for which the radiologist has included the findings of RhoTM in their report (i.e. a positively reported RhoTM screen) divided by the total number of positive RhoTM screens.
Fracture risk assessment tool (FRAX) scores | 9 months
  To compare the 10-year FRAX score as calculated using a DXA-derived T-score versus a Rho-derived T-score.

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia Oikonomou, MD, PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Holland Orthopaedic & Arthritic Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No